CLINICAL TRIAL: NCT05126927
Title: A Study to Evaluate the Safety Tolerability, Radiation Absorbed Dose,Distribution, PET Imaging and Histological Expression of 68GA-Nodaga-SNA006 in Patients With Solid Tumors.
Brief Title: A PET Imaging Agent to Assess the Level of Tumor Tissue-infiltrating CD8 + T Cells in Patients With Solid Tumors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: SmartNuclide Biopharma (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SN-2021-01
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NODAGA-SNA006 (Experimental): A PET contrast agent to assess the level of tumor tissue-infiltrating CD8 + T cells in patients with solid tumors
  Interventions: Biological: 68Ga-NODAGA-SNA006

INTERVENTIONS:
Biological: 68Ga-NODAGA-SNA006 — A PET contrast agent to assess the level of tumor tissue-infiltrating CD8 + T cells in patients with solid tumors

SUMMARY:
Primary objective To investigate the safety and tolerability profile of 68Ga- NODAGA-SNA006 in patients with solid tumors; To investigate the radiation absorbed dose characteristics of 68Ga-NODAGA-SNA006 in patients with solid tumors; To investigate the distribution profile of 68Ga-NODAGA-SNA006 in patients with solid tumors. Secondary objectives To investigate the optimal administration dose and radiation safety profile of 68Ga-NODAGA-SNA006; To investigate the PET imaging characteristics and high-quality imaging time window of 68Ga-NODAGA-SNA006 in patients with solid tumors; To explore the correlation between PET imaging characteristics of 68Ga-NODAGA-SNA006 binding to CD8 and histological CD8 expression characteristics; To explore peripheral blood T lymphocyte differentiation (CD8, CD4, CD3, etc.) in patients with solid tumors.

DETAILED DESCRIPTION:
The study had a dose-escalation, open-label design. Intravenous injection of SNA006 was used to observe its safety tolerance, radiation absorbed dose, distribution, and PET imaging characteristics in patients with solid tumors. The study consists of three phases, namely, a screening period, a trial period, and a safety follow-up period.

1. Safety evaluation Observe any AE occurred in all subjects during the clinical study, record the clinical features, severity, occurrence time, end time, duration, treatment measures and outcome, and determine the correlation between any AE and the study drug.
2. efficacy evaluation 2.1. Evaluation of imaging characteristics In this clinical trial, PET imaging characteristics will be evaluated by an independent imaging evaluation committee, and the PET imaging operating procedures and parameters will be detailed in the PET/CT standard operating procedures. 2.2. Evaluation of correlation between imaging expression and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years (including boundary values);
2. Have behavioral ability, and voluntarily participate in this clinical study, and sign the informed consent form (ICF);
3. Performance status (ECOG) score 0-1 points (see Appendix 1 for details);
4. Basal heart rate 60-100 beats/min (including boundary values);
5. Blood pressure measurement < hypertension grade 1 level (including a history of hypertension, systolic blood pressure < 140 and diastolic blood pressure < 90 mmHg by exercise or drug treatment);
6. Patients with confirmed solid tumors;
7. Patients who must have at least one image-measurable lesion according to the evaluation criteria for solid tumors (RECISTv1.1);
8. Imaging results show that at least one tumor lesion can be needle biopsy or surgical treatment to obtain specimens (enhanced CT, enhanced MRI or 18F-FDG PET/CT results are acceptable);
9. Patients with immunohistochemical CD8 results within the past month;

Exclusion Criteria:

1. Those who are unable to follow this clinical trial protocol well enough to make visits, or undergo relevant examinations, or treatment.
2. Those who have extremely poor nutritional status and cannot tolerate the trial
3. Those with comorbid major diseases or other malignancies (except those that have healed by one year or do not require additional treatment)
4. Those with known severe allergy to SNA006, similar drugs or excipients. Specialized conditions
5. Patients who have undergone previous splenectomy or splenic disease such as hypersplenism or splenomegaly
6. Patients with brain metastases.
7. Serum virology tests: positive results for any of hepatitis B virus surface antigen, hepatitis C virus antibodies, syphilis-specific antibodies or those who cannot be determined to be negative for human immunodeficiency virus antibodies
8. Patients who have not recovered from a serious infection
9. Patients with drug/alcohol abuse, severe mental disorders
10. Those with claustrophobia, emotional instability, acute persistent spasticity or inability to keep both arms up and lying flat for 15-30 minutes
11. Those who have participated in any other clinical trial within 3 months prior to screening
12. Women who are pregnant or breastfeeding.
13. Those who, in the opinion of the investigator, are not suitable to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Safety evaluation indicators | 12 months
  AE/SAE/SUSAR. To observe AE/SAE/SUSAR of subjects during trial period, until 12 months after trial finished.

SECONDARY OUTCOMES:
Immunogenicity evaluation | 1 week
  ADA blood samples were collected twice, and tested in an independent third party central laboratory. Then, ADA positive rate were analysied.
Evaluation of imaging characteristics | 12 months
  Target/background ratio in PET imaging of tumor lesions was calculated, compared target lesions with contralateral lesions, liver and muscle.
Evaluation of the correlation between imaging expression and immunohistochemistry | 12 months
  Immunohistochemical analysis (third-party independent central laboratory testing) was performed on the collected tumor tissue samples, and the scoring results were compared with the imaging expression results to calculate the sensitivity, specificity and other results.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University; Songbing Qin, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Zheng M, Zhao J, Wang C, Zhao S, Bian Y, Dai N, Zheng Y, Sang S, Guo L, Huang C, Zhang H, Jiang J, Xu C, Zhao Q, Han J, Xu T, Qin S, Miao L. Human dose-escalation study of PET imaging CD8+ T-cell infiltration in solid malignancies with [68Ga]Ga -NODAGA-SNA006. Eur J Nucl Med Mol Imaging. 2025 Mar;52(4):1332-1344. doi: 10.1007/s00259-024-06999-x. Epub 2024 Dec 10. PMID 39653817
- [Derived] Wang Y, Wang C, Huang M, Qin S, Zhao J, Sang S, Zheng M, Bian Y, Huang C, Zhang H, Guo L, Jiang J, Xu C, Dai N, Zheng Y, Han J, Yang M, Xu T, Miao L. Pilot study of a novel nanobody 68 Ga-NODAGA-SNA006 for instant PET imaging of CD8+ T cells. Eur J Nucl Med Mol Imaging. 2022 Nov;49(13):4394-4405. doi: 10.1007/s00259-022-05903-9. Epub 2022 Jul 13. PMID 35829748